CLINICAL TRIAL: NCT05422651
Title: Characteristic, Diagnosis and Prognosis of Patients Admitted With Fever in Department of Infectious Diseases
Brief Title: Observational Study About In-patients Admitted With Fever
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Huang Yan, Professor, Xiangya Hospital of Central South University
Other Study IDs: Xiangya fever project
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood includes blood cells and serum, urine and fecal samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with fever: All subjects will receive the currently recognized routine test of fever according to their disease and corresponding etiological treatment if needed and no additional intervention and treatment will be added for subjects

SUMMARY:
Fever is a common symptom in patients with infectious diseases. This study hopes to understand the epidemiological characteristics of patients hospitalized due to fever through observational research, including: clinical characteristics, etiology of fever and prognosis after treatment. So as to further search for biochemical or other serological indicators to predict the diagnosis and prognosis of infectious fever and non-infectious fever, and try to establish relevant prediction models.

DETAILED DESCRIPTION:
This study mainly prospectively analyze the clinical data of patients with fever with/without other symptoms admitted to the department of infectious diseases, Xiangya Hospital of Central South University, to analyze the epidemiological characteristics, diagnosis and prognosis of these patients. This is an observational study. All subjects will receive the currently recognized routine test of fever according to their disease and corresponding etiological treatment if needed. The researchers will collect various clinical examination indexes of the subjects in the process of diagnosis and treatment, including but not limited to white blood cells, C-reactive protein, Procalcitonin, ferritin, blood culture, therapeutic drugs, etc. Etiology and prognosis of patients will be recorded. Blood samples, urine and stool samples of all subjects will be taken after enrollment and stored for probably testing in the future. This study has no additional intervention and treatment for subjects. All subjects will sign informed consent.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to department of infectious diseases because of fever

Exclusion Criteria:

* patents who refuse to sign informed consent

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients between the age of 14-90, who were admitted to Department of Infectious Diseases because of fever with/without other symptoms were all elligible for this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Length of fever | 1 month after admission
  The interval between the onset of fever and the return of body temperature to normal after medical intervention or spontaneous remission

SECONDARY OUTCOMES:
Fever associated mortality | 3 months
  mortality of patients due to conditions associated with fever

CONTACTS AND LOCATIONS:
Overall Officials: Yan Huang, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Department of Infectious Disease, Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided